CLINICAL TRIAL: NCT00547170
Title: Efficacy and Side-Effects of Two Dosing Regimens of Doxycycline at Surgical Abortion: A Randomized Double-Blind Trial
Brief Title: Doxycycline Prophylaxis at Vacuum Aspiration Trial
Acronym: Tu Du Doxy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Tu Du Hospital (Other Government)
Responsible Party: Matthew Reeves, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO06040005
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Endometritis
Keywords: pelvic infection; abortion; doxycycline
MeSH Terms: conditions — Endometritis; Pelvic Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Half of enrolled women will be randomly assigned to group 1.
  Interventions: Drug: Doxycycline pre-operatively
- 2 (Active Comparator): Half of enrolled women will be randomly assigned to group 2
  Interventions: Drug: Doxycycline post-operatively

INTERVENTIONS:
Drug: Doxycycline pre-operatively — Two capsules of Doxycycline 100 mg before vacuum aspiration Placebo "100 mg" twice daily for 5 days after vacuum aspiration (appearance of capsules is the same for both groups)
  Arms: 1
Drug: Doxycycline post-operatively — Two capsules of placebo "100 mg" before vacuum aspiration Doxycycline 100 mg twice daily for 5 days after vacuum aspiration (appearance of capsules is the same for both groups)
  Arms: 2

SUMMARY:
This study is a randomized, double-blinded, controlled trial comparing two regimens of doxycycline for the prevention of infection after surgical abortion. One thousand women undergoing surgical abortion in the first trimester will be enrolled from the clinic at Tu Du Hospital, Ho Chi Minh City, Vietnam. The standard regimen has been 100 mg twice daily for 5 days after the abortion. Subjects will be randomized to the standard regimen or to take 200 mg doxycycline pre-operatively. Subjects found to have a positive Chlamydia EIA test will receive a 7-day course of doxycycline regardless of study group. Subjects will complete questionnaires of symptoms, including nausea and emesis in the recovery room after the procedure and at a single follow-up visit two weeks later. The primary outcome will be infection after abortion, defined below. Analyses will be performed including and excluding Chlamydia-positive subjects. Secondary outcomes will be the proportion with nausea, emesis, and other side-effects.

ELIGIBILITY:
Inclusion Criteria.

1. Women seeking elective surgical abortion
2. Gestational age 6 weeks 0 days to 12 weeks 6 days, confirmed by ultrasound.
3. Willing and able to sign an informed consent.
4. Willing to comply with the study protocol.
5. Age at enrollment of 18 years or more.

Exclusion criteria

1. Allergy to doxycycline or any tetracycline
2. Evidence of current pelvic infection
3. Breastfeeding
4. Current or recent use (within the past 7 days) of any other antibiotic.
5. Prior cardiac valve surgery or cardiac valve replacement.
6. Active use of alcohol, heroin, or cocaine.

Post-enrollment Exclusion criteria

1) Abortion procedure not performed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Infection | 2 weeks

SECONDARY OUTCOMES:
nausea and emesis | 2 weeks
compliance (completion of study medication) | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthew F Reeves, MD, Principal Investigator — University of Pittsburgh; Loi T Tran, MD, Study Director — Tu Du Hospital, Ho Chi Minh City, Vietnam
Locations (1):
- Tu Du Hospital, Ho Chi Minh City, Vietnam